CLINICAL TRIAL: NCT02007200
Title: A Phase II Trial of Preoperative Soy Isoflavone Supplementation and Molecular Markers in the Prevention of Head and Neck Squamous Carcinoma
Brief Title: Soy Isoflavones in Preventing Head and Neck Cancer Recurrence in Patients With Stage I-IV Head and Neck Cancer Undergoing Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03618; NCI-2011-03618 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UMCC 2009.008 (Other: University of Michigan Comprehensive Cancer Center); UMCC 2009.008 (Other: DCP); P30CA046592 (NIH); NCT01028001 (obsolete NCT alias)
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-09

CONDITIONS: Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Laryngeal Verrucous Carcinoma; Recurrent Lip and Oral Cavity Squamous Cell Carcinoma; Recurrent Oral Cavity Verrucous Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Stage I Hypopharyngeal Squamous Cell Carcinoma; Stage I Laryngeal Squamous Cell Carcinoma; Stage I Laryngeal Verrucous Carcinoma; Stage I Lip and Oral Cavity Squamous Cell Carcinoma; Stage I Oral Cavity Verrucous Carcinoma; Stage I Oropharyngeal Squamous Cell Carcinoma; Stage II Hypopharyngeal Squamous Cell Carcinoma; Stage II Laryngeal Squamous Cell Carcinoma; Stage II Laryngeal Verrucous Carcinoma; Stage II Lip and Oral Cavity Squamous Cell Carcinoma; Stage II Oral Cavity Verrucous Carcinoma; Stage II Oropharyngeal Squamous Cell Carcinoma; Stage III Hypopharyngeal Squamous Cell Carcinoma; Stage III Laryngeal Squamous Cell Carcinoma; Stage III Laryngeal Verrucous Carcinoma; Stage III Lip and Oral Cavity Squamous Cell Carcinoma; Stage III Oral Cavity Verrucous Carcinoma; Stage III Oropharyngeal Squamous Cell Carcinoma; Stage IV Hypopharyngeal Squamous Cell Carcinoma; Stage IVA Laryngeal Squamous Cell Carcinoma; Stage IVA Laryngeal Verrucous Carcinoma; Stage IVA Lip and Oral Cavity Squamous Cell Carcinoma; Stage IVA Oral Cavity Verrucous Carcinoma; Stage IVA Oropharyngeal Squamous Cell Carcinoma; Tongue Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lymphoid Interstitial Pneumonia; Tongue Neoplasms | interventions — Soybean Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (soy isoflavones) (Experimental): Patients receive soy isoflavones PO for approximately 14 days before undergoing surgery.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Soy Isoflavones; Other: Survey Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Soy Isoflavones — Given PO
  Other Names: NovaSoy; Solgen 40; Soy Isoflavone; Soybean Isoflavone Mixture
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase II clinical trial studies how well soy isoflavones work in preventing head and neck cancer in patients with stage I-IV head and neck cancer undergoing surgery. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of soy isoflavones may prevent head and neck cancer recurrence.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if short term, preoperative (300 mg/day x 14 treatment days) soy isoflavone supplementation modulates p16 methylation (% CpG sites methylated) and expression of p16, cyclooxygenase 2 [COX-2], vascular endothelial growth factor receptor [VEGF], epidermal growth factor receptor [EGFR], interleukin-6 [IL6], p53 and B-cell lymphoma-extra large [Bcl-xL] in tumor and non-tumor adjacent mucosa of patients with head and neck squamous carcinoma undergoing curative tumor resection.

II. To estimate correlations of tumor p16 methylation (% CpG sites methylated) with expression of p16 and levels of, IL6, VEGF, and 15-F2t-isoprostane in serum and saliva.

SECONDARY OBJECTIVES:

I. Describe the toxicity of short-term, preoperative treatment with soy isoflavone.

II. To determine overall and relapse-free survival.

OUTLINE:

Patients receive soy isoflavones orally (PO) for approximately 14 days before undergoing surgery.

After completion of treatment, patients are followed up, within the routine cancer management schedule, at 3, 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically-confirmed, resectable, squamous cell carcinoma of the oral cavity, oropharynx, larynx or hypopharynx
* Disease must be Stage I, II, III or IVa
* Tumor must be potentially surgically resectable and curable with conventional surgery and radiation therapy
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* Patients must give documented informed consent to participate in this study

Exclusion Criteria:

* Documented evidence of distant metastases
* Ongoing acute medical condition such as uncontrolled coronary artery disease, emphysema, or diabetes mellitus that would preclude surgical resection
* Pregnancy or lactation; patients of child bearing age must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of soy administration
* A medical or psychiatric illness which would compromise the patient's ability to tolerate this treatment or comply with administration of study drug
* Patients residing in prison
* Any patient with a history of breast or ovarian cancer
* Allergy to soy products

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Wolf, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (3):
- United States (3):
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Soy Isoflavones): Patients receive soy isoflavones PO for approximately 14 days before undergoing surgery.
  55 patients were enrolled. 3 of these patients did not receive treatment.
Period: Overall Study
Arm/Group | Treatment (Soy Isoflavones)
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 55 patients were enrolled. 3 patients did not undergo treatment. 13 patients had insufficient tissue and were therefore not evaluable. Only the 39 evaluable patients were included in the analysis.
Arm/Group | Treatment (Soy Isoflavones)
Number analyzed (Participants) | 39
Age, Continuous [Mean (Full Range); unit: Years] | 60 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in p16 Methylation (% CpG Sites Methylated) in Tumor Tissue After Soy Isoflavone
Description: The change in methylation will be analyzed in parallel using a linear repeated measures model. The fixed effects will be time (pre-treatment versus post-treatment), current smoking status (yes or no), their interaction, and tissue type (tumor or not). Satterthwaite's adjustment to the degrees of freedom will be applied to account for heteroscedasticity. The differential effect of soy isoflavone on tumor and non-tumor tissues between smokers and non-smokers will be assessed using linear contrasts.
Time Frame: From baseline to surgery, up to 42 days
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: Percent change
Arm/Group | Treatment (Soy Isoflavones)
Number analyzed (Participants) | 39
Percent change | 4.9 [-34.8 to 20.9]
Statistical Analysis 1: Comparison: Treatment (Soy Isoflavones); Test type: Superiority or Other; p < 0.005, Linear Repeated Measures Model

2. Primary Outcome: Correlations of Tumor p16 Methylation Status With Serum/Saliva Markers of p16, IL6, and VEGF
Description: Each of the tumor and mucosal markers will be dependent variables in repeated measures models that include serum and saliva markers as predictors. Graphical analyses will be used to characterize possible nonlinear relationships between variables. Linear or nonlinear regression, as appropriate, will be used to characterize the relationship between the putative predictors and outcomes. Subset analyses, considering, for example, differences in relationships between tumor markers and serum and saliva markers between smokers and non-smokers will be performed by means of indicator variables.
Time Frame: Up to 12 months
Population: We are seeking additional funding to hire the personnel to perform the serum/saliva markers. Until further notice markers will be unable to be analyzed.
Arm/Group | Treatment (Soy Isoflavones)
Number analyzed (Participants) | 0

3. Secondary Outcome: The Number of Participants Alive at Follow-up
Description: Overall survival at last follow-up will be determined.
Time Frame: Up to 24 months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Treatment (Soy Isoflavones)
Number analyzed (Participants) | 39
participants | 29

4. Secondary Outcome: The Number of Participants Alive Without Relapse at Last Follow-up
Description: Relapse-free survival will be determined at the last follow-up visit.
Time Frame: Up to 24 months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Treatment (Soy Isoflavones)
Number analyzed (Participants) | 39
participants | 24

ADVERSE EVENTS:
Description: 55 patients were enrolled. 3 patients did not undergo treatment. Only 52 patients were evaluable for toxicity.
Arm/Group | Treatment (Soy Isoflavones)
Serious Adverse Events (participants affected / at risk) | 7/52
Other Adverse Events (participants affected / at risk) | 25/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Soy Isoflavones) (N=52)
Cardiopulmonary arrest, cause unknown (non-fatal) (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Infection, Lung (Infections and infestations) | 1 (1)
Infection, Wound (Infections and infestations) | 1 (1)
Pain, Bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Soy Isoflavones) (N=52)
Hemoglobin (Blood and lymphatic system disorders) | 2 (24)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 3 (4)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (5)
Fever in the absence of neutropenia (General disorders) | 1 (2)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1)
Weight gain (General disorders) | 4 (5)
Weight loss (General disorders) | 3 (4)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hemorrhage, Esophagus (Vascular disorders) | 1 (1)
Hemorrhage, Oral Cavity (Vascular disorders) | 1 (1)
Infection, Blood (Infections and infestations) | 1 (1)
Infection, Neck NOS (Infections and infestations) | 1 (1)
Infection - Other (Infections and infestations) | 1 (1)
Infection, Skin (cellulitis) (Infections and infestations) | 1 (1)
Edema: head and neck (Vascular disorders) | 2 (2)
Edema: limb (Vascular disorders) | 3 (3)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 (6)
Amylase (Metabolism and nutrition disorders) | 3 (4)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 3 (4)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 6 (11)
Cholesterol, serum-high (hypercholestremia) (Metabolism and nutrition disorders) | 3 (4)
Creatinine (Metabolism and nutrition disorders) | 2 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 10 (19)
Lipase (Metabolism and nutrition disorders) | 5 (5)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 3 (6)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 5 (6)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 (7)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 (5)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (6)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 8 (10)
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint-function (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, Extraocular (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, facial (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, Whole Body (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (2)
Mood alteration, Depression (Nervous system disorders) | 1 (1)
Neurology - Other (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Pain, Abdomen NOS (Gastrointestinal disorders) | 3 (3)
Pain, Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Face (General disorders) | 1 (1)
Pain, Head (Nervous system disorders) | 1 (1)
Pain, Neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Oral (Gastrointestinal disorders) | 4 (4)
Pain, Throat (Gastrointestinal disorders) | 1 (1)
Pain - Other (General disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 2 (2)
Intra-operative injury (Surgical and medical procedures) | 1 (1)
Syndromes - Other (General disorders) | 1 (1)
Vessel injury-vein (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less